CLINICAL TRIAL: NCT05594355
Title: Effect of Treatment With EGb 761(r) on Blood Markers of Inflammation and Oxidative Stress in a Cohort of Patients With Mild Cognitive Impairment
Brief Title: Effect of Treatment With EGb 761(r) on Blood Markers of Inflammation and Oxidative Stress in Patients With MCI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fundació ACE Institut Català de Neurociències Aplicades (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACE-2020-EGb761
Record Dates: First submitted 2022-10-17; First posted 2022-10-26 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Mild Cognitive Impairment (MCI)
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): Treatment with EGb 761® (TEBOFORTAN 240 mg) during 24 months.
  Interventions: Drug: TEBOFORTAN
- Arm 2 (No Intervention): No Treatment during 12 months and treatment with EGb 761® (TEBOFORTAN 240 mg) for the next 12 months.

INTERVENTIONS:
Drug: TEBOFORTAN — TEBOFORTAN 240 mg is administrated 1 tablet per day
  Arms: Arm 1

SUMMARY:
Mild Cognitive Impairment (MCI) is the moderate impairment of a mental abilities to perform intellectual activities eg memory, calculation, communication... MCI is a disorder that can occur earlier than dementia such as Alzheimer's disease. It is believed that there are several factors involved such as inflammation and oxidative stress which is the production of reactive oxygen species that damage cells.

This clinical study tries to evaluate that a treatment already approved by the AEMPS, EGb 761® (Tebofortan), could reduce the levels of markers of inflammation and oxidation in the blood.

DETAILED DESCRIPTION:
This treatment is based on a plant called Gingko Biloba. In the study, half of the participants would be administered EGb 761® during 24 months and the other half would not receive this treatment during 12 months and will received EGb 761® for the next 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Criteria for Mild Cognitive Impairment according to Petersen.
* Global score Deterioration Scale (GDS)=3 and Clinical Dementia Rating (CDR)=0.5.
* Subject's ability to comply with study requirements in the opinion of the investigator.
* Informed consent signed

Exclusion Criteria:

* Dementia (GDS=4-7) Severe auditory or visual abnormalities that could affect performance on neuropsychological tests.
* Severe psychiatric pathology.
* Hemorrhagic diathesis or anticoagulant treatment.
* Active treatment with anticholinesterase drugs or memantine. History of epilepsy or alcoholism.
* Galactose intolerance, malabsorption of glucose or galactose.
* Previous treatment with EGb 761®.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-04-16 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Compare changes in blood marker levels of inflammation and oxidation | Between the baseline visit and follow-up visits at 6 and 12 months. All procedures in each of the visits will be carried out in a maximum period of 30 days.
  To compare the changes in the levels of blood markers of inflammation and oxidation between the baseline visit and the follow-up visits at 6 and 12 months between the study group (patients with mild cognitive impairment who receive treatment with 1 daily tablet of EGb 761® 240 mg orally) and the control group (patients with the same clinical characteristics without treatment with EGb 761®).
  Blood markers of inflammation and oxidation: in v0 (baseline), v1 (6 month), v2 (12 month). The panel of inflammation markers from Olink proteomics (https://www.olink.com/products/inflammation/) will be used with 92 proteins associated with inflammatory diseases and related biological processes. The blood samples of the participants will be collected in the Fundació ACE Nursing Unit and sent to Olink proteomics for further analysis

SECONDARY OUTCOMES:
Compare scores on neuropsychiatric tests | Between baseline visit and follow-up visit at 12 moths and follow-up visit at 24 months. All procedures in each of the visits will be carried out in a maximum period of 30 days.
  A neuropsychological evaluation will be performed in v0, v2 and v4. The neuropsychological battery may be administered in person or telematically indistinctly. Fundació ACE Battery (N-BACE) (Alegret M et al., 2012, Alegret M et al., 2013).
Compare changes in cognitive test scores | Between baseline visit, follow-up visit at 12 moths and follow-up visit at 24 months. All procedures in each of the visits will be carried out in a maximum period of 30 days.
  Neurological evaluation will be performed in v0, v2 and v4. It consists of a structured anamnesis of the patient and an informant. Data on age, sex, educational level, medical history, including cardiovascular risk factors, and treatment received are collected. A complete neurological examination using the Spanish version of the Mini Mental State Examination test is administered. Hachinski ischemia scale, the Spanish version of the Neuropsychiatric Inventory Questionnaire, the Global Deterioration Scale, the Clinical Dementia Rating and the Blessed scale.
  follow-up visit between the study group and the control group
Obtain data of changes in blood marker levels of inflammation and oxidative stress and security data | Between v0 (baseline), v1 (6 month), v2 (12 month), v3 (18 month), v4 (24 month) and in the Follow-up visit one month after the end of the treatment. All procedures in each of the visits will be carried out ina maximum period of 30 days.
  Obtain data on levels of blood markers of inflammation and oxidative stress and safety for two years in the group receiving EGb761® during the first 12 month of the study and one year in the group control.Blood markers of inflammation and oxidation: in v0 (baseline), v1 (6 month), v2 (12 month), v3 (18 month), v4 (24 month) and in the Follow-up visit one month after the end of the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Merce Rovira, MD, Principal Investigator — Fundació ACE Institut Català de Neurociències Aplicades
Locations (1):
- Fundació ACE. Institut Català de Neurociències Aplicades., Barcelona, Spain

REFERENCES:
- [Derived] Morato X, Marquie M, Tartari JP, Lafuente A, Abdelnour C, Alegret M, Jofresa S, Buendia M, Pancho A, Aguilera N, Ibarria M, Diego S, Cuevas R, Canada L, Calvet A, Antonio EE, Perez-Cordon A, Sanabria A, de Rojas I, Nunez-Llaves R, Cano A, Orellana A, Montrreal L, Canabate P, Rosende-Roca M, Vargas L, Bojaryn U, Ricciardi M, Ariton DM, Espinosa A, Ortega G, Munoz N, Lleonart N, Alarcon-Martin E, Moreno M, Preckler S, Tantinya N, Ramis M, Nogales AB, Seguer S, Martin E, Pytel V, Valero S, Gurruchaga M, Tarraga L, Ruiz A, Boada M. A randomized, open-label clinical trial in mild cognitive impairment with EGb 761 examining blood markers of inflammation and oxidative stress. Sci Rep. 2023 Apr 3;13(1):5406. doi: 10.1038/s41598-023-32515-6. PMID 37012306